CLINICAL TRIAL: NCT04436185
Title: Conducted to Determine and Compare the Effectiveness of Different Non-pharmacological Methods in Pain Management During Vaccination.
Brief Title: Effectiveness of Different Non-pharmacological Methods in Pain Management During Vaccination.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Emriye Hilal Yayan, associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: interventional
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Pain
Keywords: pain; infants
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized experimental study with placebo and control groups in order to compare the effects of ShotBlocker® and sucrose on pain reduction during vaccine injections.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the study, a multi-stage randomization method was used as follows: 1) random selection of the family health centres in the city in which the research was conducted; 2) selection of the mothers and infants to be included in the study at each centre; and 3) selection of the groups to which the participants were assigned using a computer-based block randomization method (https://www.randomizer.org). The infants, randomized via a computer system, were assigned to the ShotBlocker® group (n= 35), ShotBlocker®-placebo group (n = 35), sucrose group (n = 35), sucrose-placebo group (n = 35), or the control group (n=35).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Characteristics of newborns included (No Intervention): Characteristics of newborns included in the randomized controll
- Intraclass Correlation between the NIPS Score of Parent, Nurse (Experimental): Intraclass Correlation between the NIPS Score of Parent, Nurse
  Interventions: Behavioral: Comparisons of procedural pain
- Comparisons of procedural pain scores among groups (Experimental): Comparisons of procedural pain scores among groups
  Interventions: Behavioral: Comparisons of procedural pain

INTERVENTIONS:
Behavioral: Comparisons of procedural pain — This randomized experimental study with placebo and control groups
  Arms: Comparisons of procedural pain scores among groups; Intraclass Correlation between the NIPS Score of Parent, Nurse

SUMMARY:
Aim: This study was conducted to determine and compare the effectiveness of different non-pharmacological methods in pain management during vaccination.

Methods: This randomized experimental study with placebo and control groups was conducted with 175 infants assigned to the ShotBlocker® (n = 35), ShotBlocker®-placebo (n = 35), sucrose (n = 35), sucrose-placebo (n = 35) and control (n = 35) groups. The pain levels of the infants were determined by blind assessors (nurses, parents, and observer) using the Neonatal Infant Pain Scale (NIPS) before and during vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Born at full term
* No infection, redness, deteriorated skin integrity, or nerve damage in the area of application
* Had not undergone any clinical injection.

Exclusion Criteria:

* Infants who have applied analgesics before the vaccination

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | 10 minutes
  NIPS is a valid behavioural instrument that can be used to assess infants' response to pain. NIPS includes six behavioural responses to pain: facial expression, crying, breathing patterns, arms, legs, and state of wakefulness. The total pain scores range from 0 to 7. While the internal consistency of the original NIPS is within the range of .87 to .95, the internal consistency of the Turkish version is .83

CONTACTS AND LOCATIONS:
Locations (1):
- İnonu Üniversity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No